CLINICAL TRIAL: NCT01646606
Title: Monitoring OXYgen in Infants Hospitalized With Bronchiolitis: A Best Practices Trial (The MOXY Trial)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Sanjay Mahant, Staff Physician, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 1000029983
Record Dates: First submitted 2012-04-04; First posted 2012-07-20 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-07

CONDITIONS: Bronchiolitis
Keywords: Bronchiolitis; Length of stay; Pilot Projects; Oxygen saturation monitoring
MeSH Terms: conditions — Bronchiolitis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Continuous oxygen monitoring (Active Comparator): Oxygen saturation will be measured continuously through the child's hospital stay until discharge. Vital signs will be measured at a frequency determined by the responsible physician (as is current practice). The reading will be displayed on the bedside monitor in the participants' room.
  Interventions: Procedure: Continuous oxygen monitoring
- Intermittent oxygen monitoring (Experimental)
  Interventions: Procedure: Intermittent oxygen monitoring

INTERVENTIONS:
Procedure: Intermittent oxygen monitoring — Oxygen saturation and vital signs will be measured intermittently at a frequency of every 4 hours by the bedside nurse through the child's hospital stay until discharge. The nurse will attach the probe to the electrical cord which is connected to the monitor. For each measurement, the duration of monitoring will be until a steady wave form is present on the oxygen saturation monitor, indicating a reliable measurement (consistent with current standard of practice). The nurse will document the maximum and minimum reading during the period. The nurse will detach the probe from the electrical cord, leaving the probe attached to the child. Hence, the child's probe will be attached to the electrical cord intermittently as well.
  Arms: Intermittent oxygen monitoring
Procedure: Continuous oxygen monitoring — Oxygen saturation will be measured continuously through the child's hospital stay until discharge. Every 4 hours the nurse will complete and document a set of vital sign measurements, including oxygen saturation level, in keeping with current clinical practice. The reading will be displayed on the bedside monitor in the participants' room. At the completion of vital signs measurement, the nurse will not detach the electrical cord from the probe. Hence, the child's probe will be attached to the electrical cord continuously as well.
  Arms: Continuous oxygen monitoring

SUMMARY:
In infants hospitalized with bronchiolitis, a common infection in the lungs caused by a virus, it is uncertain on how to best monitor their oxygen levels. It is common to place a probe on infants hands or legs to monitor oxygen levels. The probe can be used to monitor oxygen levels all the time (continuous oxygen monitoring) or just every 4-6 hours (intermittent oxygen monitoring). There is reason to believe that placing children with bronchiolitis on continuous monitoring might result in children staying longer in hospital than needed. This is a research study that is aiming to provide data to plan a larger research study to answer the question of whether intermittent oxygen monitoring is better than continuous oxygen monitoring. This study is part of a larger initiative to determine the best way to care for children with bronchiolitis, including making sure that children do not stay in hospital longer than needed.

Parents will be asked to participate in this research study if their child is hospitalized with bronchiolitis and has been stable for at least 6 hours, meaning that he/she is not having more trouble breathing or does not require more supplemental oxygen. If they agree participate, the child will have one of the two oxygen monitoring strategies: intermittent or continuous monitoring. Each child will have an equal chance of getting one or the other of these two monitoring strategies.

The study team will review the children's charts to determine the number of tests ordered, the need for intensive care unit help or admissions, the number of blood tests and chest x-rays the treating doctors ordered, and the length of hospital stay. Parents will be contacted about 4-5 days after discharge to ask if there were any unscheduled visits to doctors or emergency rooms after discharge. The investigators will the parents to fill out a scale twice a day asking how well their child is feeding. The investigators will also them to rate their anxiety level once a day.

The information from this study will help plan and support an application for external funding. The results of a larger study could potentially decrease unnecessary monitoring, oxygen supplementation, and hospital stay and thereby improve quality of care with large cost savings. A reduction in length of hospital stay for this common hospital condition would also reduce the burden of hospitalization to families and reduce the risks associated with harm in the hospital setting such as infection and medical error.

ELIGIBILITY:
Inclusion Criteria:

* First episode of acute bronchiolitis.
* Clinical diagnosis of bronchiolitis as defined by the American Academic of Pediatrics Clinical Practice Guideline: Diagnosis and Management of Bronchiolitis as a constellation of clinical findings on history and physical exam; clinical findings include 1) a preceding viral upper respiratory infection; 2) presence of wheeze on chest auscultation; 3) increased respiratory effort
* Clinical status stable for 6 hours as defined by 1) stable or decreasing requirement for supplemental oxygen AND a stable or decreasing respiratory rate (within 10 breaths per minute) on at least two measurements; 2) respiratory rate < 70 breaths/minute; 3) oxygen supplementation < 40% FiO2 or < 2 L/min by nasal prongs; and 4) heart rate < 180 beats per minute
* Availability of home telephone or mobile cell phone to contact the participant's parent/guardian after discharge from hospital

Exclusion Criteria:

* Preexisting chronic medical condition which includes the following: 1) congenital heart disease that is cyanotic, hemodynamically significant requiring diuretics, and/or with pulmonary hypertension; 2) chronic lung disease with home oxygen requirement and/or pulmonary hypertension; 3)neuromuscular disease; 4) immunodeficiency; or 5) hemoglobinopathy
* Premature birth (< 36 weeks)
* History of apnea on current admission
* Receiving morphine infusions
* Weight < 4kg

Ages: 6 Weeks to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 33 (Actual)
Dates: Start 2012-03; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Length of hospital stay | Admission - Discharge (up to 2 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay Mahant, MD, MSc, Principal Investigator — The Hospital for Sick Children
Locations (1):
- Hospital for Sick Children, Toronto, Ontario, Canada